CLINICAL TRIAL: NCT06744218
Title: Effectiveness of Telerehabilitation as an Alternative to Outpatient Physiotherapy in the 1 Month After Arthroscopic Rotator Cuff Repair Surgery: Multicenter Randomized Clinical Trial
Brief Title: Effectiveness of Telerehabilitation as an Alternative to Outpatient Physiotherapy in the 1 Month After Arthroscopic Rotator Cuff Repair Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Teleriab-Cuffia
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Injuries
Keywords: telerehabilitation; physiotherapist; rotator cuff repair surgery
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator)
  Interventions: Procedure: Standard Treatment
- experimental (Experimental)
  Interventions: Procedure: Experimental Treatment

INTERVENTIONS:
Procedure: Standard Treatment — Patients who will be assigned to the control group and subjected to standard treatment (usual care at our clinic) will undergo a physiotherapy treatment of 8 in-person sessions for 4 post-operative weeks
  Arms: Standard
Procedure: Experimental Treatment — patients who will be assigned to the experimental group and subjected to the experimental treatment will undergo a physiotherapy treatment of 8 sessions in telerehabilitation for 4 post-operative weeks
  Arms: experimental

SUMMARY:
The present study aims to verify whether telerehabilitation as an alternative to in-person treatment (both conducted by a physiotherapist) can be a valid option in terms of pain, recovery of the rom, shoulder functionality compared to those provided by therapy alone. face-to-face rehabilitation in patients undergoing arthroscopic rotator cuff repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 40 and 70 years
* Patients undergoing arthroscopic repair surgery of the rotator cuff tendons
* Start of outpatient treatment within 7 days of discharge from the Orthopedic Department of the Argenta and Delta hospitals
* Continuation of rehabilitation care at the IOR Physical and Rehabilitation Medicine service in Argenta or at the Physical Therapy Rehabilitation Medicine service of the Delta Hospital.
* Patients who have provided informed consent

Exclusion Criteria:

* Previous shoulder surgeries
* difficulty understanding the Italian language/language barrier
* unavailability of IT devices or stable wi-fi connection by the patient

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Score | At baseline (day 0), after one months, after 3 months
  The Constant-Murley score (CMS) is a 100-point scale made up of a series of individual parameters. These parameters define the patient's pain level and ability to carry out normal daily activities

SECONDARY OUTCOMES:
Mobility of the shoulder | At baseline (day 0), after one months, after 3 months
  Range of motion of the shoulder seen by movements made during the rehabilitation
Numeric rating scale | At baseline (day 0), after one months, after 3 months
  Description of pain by numeric rating scale, from 0 no pain, to 10 worst pain ever (0-10)
Disabilities of the Arm, Shoulder and Hand | at baseline, after 3 months and after 6 months
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that examines a patient's ability to perform certain upper extremity activities

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale del Delta, Lagosanto, Ferrara
  - IRCCS Istituto ortopedico Rizzoli, Bologna, Italia